CLINICAL TRIAL: NCT01887912
Title: Efficacy, Immunogenicity, and Safety Study of Clostridium Difficile Toxoid Vaccine in Subjects at Risk for C. Difficile Infection (Cdiffense™)
Brief Title: Study of a Candidate Clostridium Difficile Toxoid Vaccine in Subjects at Risk for C. Difficile Infection
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The Independent Data Monitoring Committee (IDMC) concluded that the probability that the study will meet its primary objective is low.
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H-030-014; 2013-000775-32 (EudraCT Number); U1111-1127-7162 (Other: WHO)
Record Dates: First submitted 2013-06-20; First posted 2013-06-27 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Clostridium Difficile Infection
Keywords: Clostridium difficile Toxoid Vaccine; Clostridium difficile infection; Cdiffense
MeSH Terms: conditions — Clostridium Infections | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: This study was observer-blind. The vaccine preparer and administrator may have been unblinded to treatment assignment due to the steps necessary for vaccine preparation. However, the participant, the Investigator, and study staff members who collected the safety data and laboratory personnel who analyzed the blood and stool samples were all blinded to the group assignment.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- C. difficile Vaccine Group (Experimental): Participants received 1 injection of 0.5 mL C. difficile toxoid vaccine at Days 0 (Injection 1), 7 (Injection 2), and 30 (Injection 3).
  Interventions: Biological: C. difficile Toxoid Vaccine
- Placebo Group (Placebo Comparator): Participants received 1 injection of 0.5 mL placebo matched to vaccine at Days 0 (Injection 1), 7 (Injection 2), and 30 (Injection 3).
  Interventions: Biological: Placebo: 0.9% normal saline

INTERVENTIONS:
Biological: C. difficile Toxoid Vaccine — 0.5 mL, Intramuscular
  Arms: C. difficile Vaccine Group
Biological: Placebo: 0.9% normal saline — 0.5 mL, Intramuscular
  Arms: Placebo Group

SUMMARY:
The aim of this study was to evaluate the efficacy of the Clostridium difficile vaccine to prevent primary symptomatic C. difficile infection (CDI) in participants at risk for CDI where there is a substantial unmet medical need.

Primary objective:

* To assess the efficacy of the C. difficile vaccine in preventing the onset of symptomatic primary CDI confirmed by polymerase chain reaction (PCR) in adult participants aged >= 50 years who are at risk for CDI and have received at least 1 injection.

Secondary Objectives:

Efficacy:

* To assess prevention of symptomatic PCR-confirmed primary CDI cases after 3 injections administered at 0, 7, and 30 days.
* To assess prevention of symptomatic PCR-confirmed primary CDI cases after completion of at least 2 injections.

Immunogenicity:

* To describe the immunogenicity to toxin A and toxin B at specific time points in a subset of participant and in participants with CDI at Day 0 and Day 60.

Safety:

* To describe the safety profile of all participants who received at least 1 injection.

DETAILED DESCRIPTION:
The study was designed as an event-driven group sequential protocol with 4 interim analyses at defined information milestones and a final analysis when a specific number of clinical endpoints are reached. Analyses of trial futility (non-efficacy) were to be performed at the first 2 interim analyses, and the study was to be stopped if either of those analyses provided robust and compelling evidence that meaningful levels of vaccine efficacy (VE) would not be demonstrated.

Following completion of the first interim analysis (50 cases of confirmed CDI observed), the futility criterion was met and in accordance with IDMC recommendation, enrollment and further vaccination ceased in November 2017.

Due to the early termination of the study, some of the planned secondary efficacy endpoints could not be analyzed as all planned data were not collected.

Participants were randomized to receive either the candidate vaccine or a placebo that was to be administered in a 3-dose schedule. At the time of group assignment, 928 participants (10% of total enrollment) were randomized to an immunogenicity subset; and 1859 participants (20% of total enrollment) were randomized to a reactogenicity subset.

Safety was assessed in all participants in terms of unsolicited adverse events from Day 0 to Day 60, as well as serious adverse events (SAEs) throughout the study. Solicited adverse reactions were collected for 6 days following each injection in the reactogenicity subset.

ELIGIBILITY:
Inclusion Criteria:

* Aged >= 50 years on the day of inclusion
* Informed consent form had been signed and dated.
* Attended all scheduled visits and complied with all trial procedures.
* Covered by health insurance (if required).
* Must fulfill at least 1 of the following criteria

Risk Stratum 1:

* Had at least 2 hospital stays, each lasting at least >= 24 hours, in the 12 months before enrollment, and
* Had received systemic (not topical) antibiotics in the 12 months before enrollment, or

Risk Stratum 2:

* Was anticipated to have an in-patient hospitalization for a planned surgical procedure within 60 days of enrollment. The impending hospital stay was planned to be >= 72 hours for a surgery involving 1 of the following:
* Kidney/bladder/urinary system
* Musculoskeletal system
* Respiratory system
* Circulatory system
* Central nervous system.

Exclusion Criteria:

* Participant was pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be post-menopausal for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination and until at least 4 weeks after the last vaccination).
* Participation in the 4 weeks preceding the first trial vaccination or participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination except for influenza (seasonal or pandemic) and pneumococcal vaccines. This exception includes monovalent pandemic influenza vaccines and multivalent influenza vaccines.
* Previous vaccination against C. difficile with either the trial vaccine, another vaccine, or monoclonal antibodies.
* Diarrhea on day of enrollment.
* Self-reported current or prior CDI episode.
* Anticipated or current receipt of kidney dialysis treatment.
* History of gastrointestinal surgery for gastrointestinal malignancy (Note: Colonoscopy, polypectomy, and appendectomy are not exclusion criteria).
* History of inflammatory bowel disease, irritable bowel syndrome (must include diarrhea as a symptom), colostomy, or small or large intestine bowel surgery where resection was performed.
* Receiving enteral feeding (e.g., nasogastric, gastrostomy, and jejunostomy tube feeding).
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the trial or to a vaccine containing any of the same substances.
* Self-reported thrombocytopenia, contraindicating intramuscular vaccination.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol abuse or drug addiction that might interfere with the ability to comply with trial procedures in the opinion of the Investigator.
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion.
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature >= 38.0 degree Celsius [>= 100.4°Fahrenheit]). A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9302 (Actual)
Dates: Start 2013-07-30 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (320):
- United States (134):
  - Huntsville, Alabama
  - Investigational Site 104, Mobile, Alabama
  - Flagstaff, Arizona
  - Investigational Site 194, Phoenix, Arizona
  - Investigational Site 503, Surprise, Arizona
  - Little Rock, Arkansas
  - Bakersfield, California
  - Banning, California
  - Garden Grove, California
  - La Mesa, California
  - Investigational Site 534, Los Angeles, California
  - Investigational Site 051, Los Angeles, California
  - Modesto, California
  - Redding, California
  - Sacramento, California
  - Investigational Site 504, Simi Valley, California
  - Investigational Site 057, Stanford, California
  - Investigational Site 176, Upland, California
  - Ventura, California
  - Investigational Site 546, Wheat Ridge, Colorado
  - Bristol, Connecticut
  - Danbury, Connecticut
  - Investigational Site 143, Bradenton, Florida
  - Investigational Site 187, Brandon, Florida
  - Investigational Site 075, Clearwater, Florida
  - Investigational Site 517, Clearwater, Florida
  - Investigational Site 055, Crystal River, Florida
  - DeLand, Florida
  - Investigational Site 506, Gainesville, Florida
  - Investigational Site 099, Hialeah, Florida
  - Investigational Site 009, Jacksonville, Florida
  - Lauderdale Lakes, Florida
  - Miami, Florida
  - Orange Park, Florida
  - Investigational Site 112, Pensacola, Florida
  - Port Saint Lucie, Florida
  - Investigational Site 088, Sarasota, Florida
  - Investigational Site 040, St. Petersburg, Florida
  - Investigational Site 114, St. Petersburg, Florida
  - Tamarac, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Investigational Site 149, Augusta, Georgia
  - Investigational Site 529, Decatur, Georgia
  - Macon, Georgia
  - Investigational Site 010, Savannah, Georgia
  - Investigational Site 049, Idaho Falls, Idaho
  - Investigational Site 543, Pocatello, Idaho
  - Evanston, Illinois
  - Peoria, Illinois
  - Anderson, Indiana
  - Investigational Site 101, Iowa City, Iowa
  - Topeka, Kansas
  - Louisville, Kentucky
  - Investigational Site 091, Metairie, Louisiana
  - Investigational Site 084, New Orleans, Louisiana
  - Opelousas, Louisiana
  - Investigational Site 077, Shreveport, Louisiana
  - Auburn, Maine
  - Baltimore, Maryland
  - Investigational Site 002, Boston, Massachusetts
  - Investigational Site 035, West Roxbury, Massachusetts
  - Investigational Site 190, Ann Arbor, Michigan
  - Investigational Site 175, Detroit, Michigan
  - Investigational Site 183, Flint, Michigan
  - Grosse Pointe Woods, Michigan
  - Kalamazoo, Michigan
  - Livonia, Michigan
  - Investigational Site 069, Royal Oak, Michigan
  - Stevensville, Michigan
  - Troy, Michigan
  - Butte, Montana
  - Investigational Site 189, Hillsborough, New Jersey
  - Investigational Site 044, Neptune City, New Jersey
  - Teaneck, New Jersey
  - Albuquerque, New Mexico
  - Investigational Site 022, Endwell, New York
  - Rochester, New York
  - Syracuse, New York
  - The Bronx, New York
  - Investigational Site 013, The Bronx, New York
  - Investigational Site 146, Asheville, North Carolina
  - Cary, North Carolina
  - Charlotte, North Carolina
  - Hickory, North Carolina
  - Raleigh, North Carolina
  - Statesville, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Investigational Site 031, Fargo, North Dakota
  - Fargo, North Dakota
  - Investigational Site 523, Canton, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Investigational Site 129, Cleveland, Ohio
  - Investigational Site 003, Columbus, Ohio
  - Investigational Site 061, Dayton, Ohio
  - Dayton, Ohio
  - Kettering, Ohio
  - Marion, Ohio
  - Investigational Site 095, Middletown, Ohio
  - Bend, Oregon
  - Investigational Site 528, Camp Hill, Pennsylvania
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Investigational Site 083, Uniontown, Pennsylvania
  - West Reading, Pennsylvania
  - Investigational Site 020, Wilkes-Barre, Pennsylvania
  - Investigational Site 050, Pawtucket, Rhode Island
  - Providence, Rhode Island
  - Investigational Site 540, Charleston, South Carolina
  - Investigational Site 047, Mt. Pleasant, South Carolina
  - Investigational Site 180, Spartanburg, South Carolina
  - Investigational Site 086, Rapid City, South Dakota
  - Franklin, Tennessee
  - Jackson, Tennessee
  - Nashville, Tennessee
  - Investigational Site 544, Austin, Texas
  - Corpus Christi, Texas
  - Investigational Site 006, Dallas, Texas
  - Investigational Site 119, Fort Worth, Texas
  - Groesbeck, Texas
  - Investigational Site 193, San Antonio, Texas
  - Tomball, Texas
  - Investigational Site 135, Orem, Utah
  - Investigational Site 080, Salt Lake City, Utah
  - Investigational Site 012, Lynchburg, Virginia
  - Williamsburg, Virginia
  - Investigational Site 196, Winchester, Virginia
  - Spokane, Washington
  - Tacoma, Washington
  - Investigational Site 030, Marshfield, Wisconsin
  - Weston, Wisconsin
- Australia (7):
  - Westmead, New South Wales
  - Investigational Site 401, Cairns, Queensland
  - Woolloongabba, Queensland
  - Investigational Site 404, Bedford Park, South Australia
  - Investigational Site 403, Clayton, Victoria
  - Nedlands, Western Australia
  - Subiaco, Western Australia
- Brazil (13):
  - Salvador, Estado de Bahia
  - Aparecida de Goiânia, Goiás
  - Belo Horizonte, Minas Gerais
  - Juiz de Fora, Minas Gerais
  - Curitiba, Paraná
  - Recife, Pernambuco
  - Nova Iguaçu, Rio de Janeiro
  - Rio de Janeiro, Rio de Janeiro
  - Natal, Rio Grande do Norte
  - Canoas, Rio Grande do Sul
  - Porto Alegre, Rio Grande do Sul
  - Santo André, São Paulo
  - Campinas
- Canada (13):
  - New Westminster, British Columbia
  - Investigational Site 156, Surrey, British Columbia
  - Investigational Site 158, Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Halifax, Nova Scotia
  - Investigational Site 163, Truro, Nova Scotia
  - Guelph, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Pierrefonds, Quebec
  - Investigational Site 152, Québec, Quebec
  - Investigational Site 151, Sherbrooke, Quebec
  - Investigational Site 161, Trois-Rivières, Quebec
- Colombia (8):
  - Barranquilla, Alantico
  - Medellín, Antioquia
  - Bogotá, Ditrito Capital
  - Bogotá, Ditrito
  - Armenia, Quindío Department
  - Bucaramanga, Santander Department
  - Floridablanca, Santander Department
  - Yopal
- San José, Costa Rica
- Investigational Site 215, Aarhus, Denmark
- Investigational Site 347, Santo Domingo, Dominican Republic
- Finland (10):
  - Espoo
  - Helsinki
  - Investigational Site 203, Jarvenpaa
  - Kokkola
  - Oulu
  - Pori
  - Seinäjoki
  - Investigational Site 201, Tampere
  - Investigational Site 202, Turku
  - Vantaa
- France (12):
  - Investigational Site 230, Dijon
  - Lille
  - Limoges
  - Lyon
  - Montpellier
  - Orléans
  - Investigational Site 221, Paris
  - Investigational Site 229, Pringy
  - Saint-Etienne
  - Investigational Site 223, Saint-Priest-en-Jarez
  - Tourcoing
  - Investigational Site 232, Tours
- Germany (12):
  - Investigational Site 244, Deggingen, Baden-Wurttemberg
  - Munich, Bavaria
  - Investigational Site 242, Würzburg, Bavaria
  - Cologne, North Rhine-Westphalia
  - Leipzig, Saxony
  - Jena, Thuringia
  - Berlin
  - Essen
  - Goch
  - Investigational Site 247, Hamburg
  - Investigational Site 245, Hamburg
  - Leipzig
- Guatemala City, Guatemala
- Japan (20):
  - Investigational Site 450, Aichi
  - Investigational Site 468, Chiba
  - Investigational Site 467, Fukui
  - Investigational Site 464, Fukuoka
  - Investigational Site 465, Fukuoka
  - Investigational Site 466, Fukuoka
  - Investigational Site 457, Gunma
  - Investigational Site 455, Hyōgo
  - Investigational Site 453, Ibaraki
  - Investigational Site 460, Kyoto
  - Investigational Site 454, Kyoto
  - Investigational Site 456, Nagano
  - Investigational Site 452, Nagano
  - Investigational Site 458, Nagano
  - Investigational Site 469, Okinawa
  - Investigational Site 461, Ōsaka
  - Investigational Site 459, Saitama
  - Investigational Site 467, Shimonoseki
  - Investigational Site 451, Tokyo
  - Investigational Site 463, Yamaguchi
- Mexico (13):
  - Aguascalientes, Aguascalientes
  - Investigational Site 325, Mexico City, D.F.
  - Investigational Site 329, Mexico City, D.F.
  - Tijuana, Estado de Baja California
  - Investigational Site 324, Guadalajara, Jalisco
  - Investigational Site 351, Cuernavaca, Morelos
  - Monterrey, Nuevo León
  - San Luis Potosí City, San Luis Potosí
  - Investigational Site 352, Ecatepec de Morelos, State of Mexico
  - Investigational Site 363, Ciudad Victoria, Tamaulipas
  - Investigational Site 326, Durango
  - Morelos
  - San Luis Potosí City
- Investigational Site 354, Panama City, Panama
- Peru (9):
  - Investigational Site 364, Trujillo, La Libertad
  - Investigational Site 332, Jesus Maria, Lima region
  - Lima Cercado, Lima region
  - Investigational Site 334, San Martín de Porres, Lima region
  - Surquillo, Lima region
  - Investigational Site 356, Lima
  - Investigational Site 355, Lima
  - Lima
  - Investigational Site 365, Piura
- Philippines (5):
  - Alabang
  - Dasmariñas
  - Manila
  - Pasig
  - Quezon City
- Poland (2):
  - Investigational Site 284, Bydgoszcz
  - Investigational Site 283, Nowy Duninów
- Puerto Rico (2):
  - Investigational Site 171, Bayamón, PR
  - Bayamón
- Singapore (4):
  - Singapore
  - Investigational Site 419, Singapore
  - Investigational Site 428, Singapore
  - Investigational Site 445, Singapore
- South Korea (22):
  - Seoul, Gangnam-gu
  - Investigational Site 407, Wŏnju, Gangwon-do
  - Investigational Site 413, Ansan, Gyeonggi-do
  - Daegu, Jung-Gu
  - Investigational Site 427, Incheon, Namdong-gu
  - Seoul, Seocho-gu
  - Seoul, Seodaemun-gu
  - Seoul, Seongbuk-gu
  - Seoul, Seongdong-gu
  - Seoul, Songpa-gu
  - Investigational Site 446, Busan
  - Cheongju-si
  - Investigational Site 439, Gyeonggi-do
  - Gyeonggi-do
  - Investigational Site 412, Incheon
  - Investigational Site 409, Seoul
  - Investigational Site 408, Seoul
  - Investigational Site 415, Seoul
  - Investigational Site 418, Seoul
  - Investigational Site 411, Seoul
  - Investigational Site 437, Seoul
  - Investigational Site 438, Seoul
- Spain (4):
  - Investigational Site 294, Córdoba
  - Investigational Site 293, Santander
  - Investigational Site 292, Terrassa
  - Investigational Site 295, Vigo
- Sweden (3):
  - Göthenburg, SWE
  - Stockholm
  - Umeå
- Taiwan (7):
  - Kaohsiung City
  - Investigational Site 426, New Taipei City
  - New Taipei City
  - Investigational Site 429, Taichung
  - Investigational Site 421, Tainan
  - Investigational Site 425, Taipei
  - Tiachung
- Thailand (3):
  - Investigational Site 443, Bangkok
  - Investigational Site 442, Bangkok
  - Investigational Site 441, Khon Kaen
- United Kingdom (12):
  - Investigational Site 276, Blackpool
  - Blackpool
  - Investigational Site 277, Coventry
  - Harrow
  - Investigational Site 281, Leeds
  - Liverpool
  - Investigational Site 271, London
  - Manchester
  - Middlesex
  - North Shields
  - Investigational Site 275, Penzance
  - Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] de Bruyn G, Gordon DL, Steiner T, Tambyah P, Cosgrove C, Martens M, Bassily E, Chan ES, Patel D, Chen J, Torre-Cisneros J, Fernando De Magalhaes Francesconi C, Gesser R, Jeanfreau R, Launay O, Laot T, Morfin-Otero R, Oviedo-Orta E, Park YS, Piazza FM, Rehm C, Rivas E, Self S, Gurunathan S. Safety, immunogenicity, and efficacy of a Clostridioides difficile toxoid vaccine candidate: a phase 3 multicentre, observer-blind, randomised, controlled trial. Lancet Infect Dis. 2021 Feb;21(2):252-262. doi: 10.1016/S1473-3099(20)30331-5. Epub 2020 Sep 15. PMID 32946836

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled in the study from 30 July 2013 to 17 November 2017.
Pre-assignment Details: A total of 9302 participants were enrolled and randomized in the study.
Period: Overall Study
Arm/Group | C. Difficile Vaccine Group | Placebo Group
Started | 6201 | 3101
Safety Population (Participants who had received the study or control vaccine, analyzed according to vaccine received) | 6113 | 3057
Completed | 4809 | 2370
Not Completed | 1392 | 731
Not completed — Serious adverse event | 400 | 198
Not completed — Other Adverse Event | 34 | 15
Not completed — Protocol Violation | 67 | 37
Not completed — Lost to Follow-up | 163 | 74
Not completed — Withdrawal by Subject | 606 | 349
Not completed — Other | 122 | 58

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | C. Difficile Vaccine Group | Placebo Group | Total
Number analyzed (Participants) | 6201 | 3101 | 9302
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (8.86) | 65.8 (8.87) | 65.8 (8.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2629 | 1294 | 3923
  Male | 3572 | 1807 | 5379
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 330 | 171 | 501
  Not Hispanic or Latino | 2780 | 1390 | 4170
  Unknown or Not Reported | 3091 | 1540 | 4631
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 6 | 12
  Asian | 795 | 398 | 1193
  Native Hawaiian or Other Pacific Islander | 5 | 4 | 9
  Black or African American | 206 | 102 | 308
  White | 2983 | 1487 | 4470
  More than one race | 8 | 5 | 13
  Unknown or Not Reported | 2198 | 1099 | 3297

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Symptomatic Polymerase Chain Reaction (PCR)-Confirmed Primary C. Difficile Infection (CDI) Cases
Description: Symptomatic PCR-confirmed CDI cases were defined as the number of participants with combination of clinical and laboratory findings. Clinical components were: >= 3 loose stools in <= 24 hours, loose stools (defined as type 6 [fluffy pieces with ragged edges, mushy] or type 7 [watery, no solid pieces] according to the Bristol Stool Chart) lasting >= 24 hours. Laboratory findings were: stool sample positive for C. difficile Toxin B by PCR at central laboratory or diagnosis of pseudomembranous colitis visualized at colonoscopy.
Time Frame: Up to 3 years post injection 1
Population: Analysis was performed on modified intent-to-treat (mITT) population which included all participants who received at least 1 injection and were analyzed according to the group to which they were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | C. Difficile Vaccine Group | Placebo Group
Number analyzed (Participants) | 6173 | 3085
Participants | 34 | 16

2. Secondary Outcome: Number of Participants With Severe PCR-Confirmed Primary CDI Cases
Description: Severe CDI cases were defined as number of participants with at least one of the following symptoms: fever >= 38.5 degree Celsius (°C), white blood cell count >= 15,000 cells/mm^3, ileus, pseudomembranous colitis, serum albumin <3 gram per deciliter, abdominal distension, abdominal tenderness, or admission to the intensive care unit within 7 days of CDI diagnosis.
Time Frame: Up to 3 years post injection 1
Population: Analysis was performed on participants with protocol-defined (PCR confirmed) primary CDI cases.
Measure: Count of Participants; unit: Participants
Arm/Group | C. Difficile Vaccine Group | Placebo Group
Number analyzed (Participants) | 34 | 16
Participants | 9 | 6

3. Secondary Outcome: Number of Participants With Loose Stool Episodes
Description: Loose stools were defined as type 6 (fluffy pieces with ragged edges, mushy) or type 7 (watery, no solid pieces) according to the Bristol Stool Chart. In this outcome measure, participants with number of loose stool episodes (categorized as: loose stool episodes less than 3, 3 to 6, 7 to 10, 11 to 15 and greater than 15) were reported.
Time Frame: Up to 3 years post injection 1
Population: Analysis was performed on participants with protocol-defined PCR confirmed CDI cases.
Measure: Count of Participants; unit: Participants
Arm/Group | C. Difficile Vaccine Group | Placebo Group
Number analyzed (Participants) | 34 | 16
Participants
  <3 | 0 | 0
  3 to 6 | 7 | 4
  7 to 10 | 7 | 2
  11 to 15 | 7 | 4
  >15 | 13 | 6

4. Secondary Outcome: Number of Participants With Symptomatic PCR Confirmed CDI Cases: Per-Protocol Population
Description: Symptomatic PCR confirmed CDI cases were defined as the number of participants with combination of clinical and laboratory findings. Clinical components were: >= 3 loose stools in <= 24 hours, loose stools (defined as type 6 [fluffy pieces with ragged edges, mushy] or type 7 [watery, no solid pieces] according to the Bristol Stool Chart) lasting >= 24 hours. Laboratory findings were: stool sample positive for C. difficile Toxin B by PCR at central laboratory or diagnosis of pseudomembranous colitis visualized at colonoscopy. Analysis was performed on per-protocol efficacy analysis set (PPEAS).
Time Frame: Up to 3 years post injection 1
Population: PPEAS: participants who had at least 1 injection, no relevant protocol deviations (not meet inclusion criteria/ met exclusion criteria, not receive any vaccine/not received in proper time window, received different vaccine than randomized, preparation and / or administration of vaccine not done per protocol, received protocol-restricted therapy).
Measure: Count of Participants; unit: Participants
Arm/Group | C. Difficile Vaccine Group | Placebo Group
Number analyzed (Participants) | 4786 | 2378
Participants | 23 | 13

5. Secondary Outcome: Serum Antibody Concentrations Against Toxins A and B Measured by Enzyme-Linked Immunosorbent Assay (ELISA)
Description: Serum antibody concentrations against toxins A and B were measured by ELISA and expressed as geometric mean concentration (GMC). The 2-sided 95% Confidence Interval (CI) of GMC was based on the Student t-distribution. Analysis was performed on Per Protocol Immunogenicity Analysis Set, which included participants who had at least 1 injection, no relevant protocol deviations (not met inclusion criteria/ met exclusion criteria, not received vaccine/ not received in proper time window, received different vaccine than randomized, preparation and/ or administration of vaccine not per protocol, protocol-restricted therapy, not provided post-dose serology sample/serology sample did not produced a valid test result).
Time Frame: Day 0, Day 14, Day 30, Day 60, Day 210, Day 390, Day 570, Day 750, Day 930, and Day 1110
Population: Analysis was performed on Per Protocol Immunogenicity Analysis Set. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units per milliliter (EU/mL)
Arm/Group | C. Difficile Vaccine Group | Placebo Group
Number analyzed (Participants) | 471 | 236
ELISA units per milliliter (EU/mL)
  Toxin A ImunnoglobulinG (IgG): Day 0: number analyzed (Participants) | 468 | 230
  Toxin A ImunnoglobulinG (IgG): Day 0 | 0.957 [0.897 to 1.02] | 0.999 [0.912 to 1.09]
  Toxin A IgG: Day 14: number analyzed (Participants) | 418 | 214
  Toxin A IgG: Day 14 | 3.19 [2.68 to 3.80] | 0.913 [0.849 to 0.983]
  Toxin A IgG: Day 30: number analyzed (Participants) | 456 | 230
  Toxin A IgG: Day 30 | 12.2 [10.4 to 14.3] | 0.959 [0.889 to 1.03]
  Toxin A IgG: Day 60: number analyzed (Participants) | 417 | 212
  Toxin A IgG: Day 60 | 43.7 [38.1 to 50.2] | 0.933 [0.867 to 1.00]
  Toxin A IgG: Day 210: number analyzed (Participants) | 355 | 182
  Toxin A IgG: Day 210 | 12.0 [10.5 to 13.8] | 0.944 [0.865 to 1.03]
  Toxin A IgG: Day 390: number analyzed (Participants) | 320 | 159
  Toxin A IgG: Day 390 | 6.02 [5.23 to 6.93] | 0.955 [0.856 to 1.06]
  Toxin A IgG: Day 570: number analyzed (Participants) | 277 | 145
  Toxin A IgG: Day 570 | 4.50 [3.86 to 5.25] | 0.908 [0.834 to 0.989]
  Toxin A IgG: Day 750: number analyzed (Participants) | 191 | 93
  Toxin A IgG: Day 750 | 4.02 [3.38 to 4.78] | 0.856 [0.776 to 0.944]
  Toxin A IgG: Day 930: number analyzed (Participants) | 108 | 66
  Toxin A IgG: Day 930 | 3.83 [3.02 to 4.85] | 0.902 [0.796 to 1.02]
  Toxin A IgG: Day 1110: number analyzed (Participants) | 59 | 36
  Toxin A IgG: Day 1110 | 3.75 [2.64 to 5.34] | 1.09 [0.786 to 1.50]
  Toxin B IgG: Day 0: number analyzed (Participants) | 468 | 231
  Toxin B IgG: Day 0 | 1.40 [1.24 to 1.57] | 1.49 [1.24 to 1.79]
  Toxin B IgG: Day 14: number analyzed (Participants) | 419 | 216
  Toxin B IgG: Day 14 | 4.36 [3.37 to 5.64] | 1.56 [1.29 to 1.89]
  Toxin B IgG: Day 30: number analyzed (Participants) | 455 | 231
  Toxin B IgG: Day 30 | 10.0 [7.85 to 12.8] | 1.46 [1.21 to 1.75]
  Toxin B IgG: Day 60: number analyzed (Participants) | 417 | 212
  Toxin B IgG: Day 60 | 24.8 [20.1 to 30.6] | 1.42 [1.18 to 1.71]
  Toxin B IgG: Day 210: number analyzed (Participants) | 354 | 182
  Toxin B IgG: Day 210 | 6.62 [5.36 to 8.19] | 1.31 [1.07 to 1.61]
  Toxin B IgG: Day 390: number analyzed (Participants) | 319 | 159
  Toxin B IgG: Day 390 | 3.98 [3.15 to 5.02] | 1.24 [0.991 to 1.56]
  Toxin B IgG: Day 570: number analyzed (Participants) | 277 | 145
  Toxin B IgG: Day 570 | 3.37 [2.63 to 4.32] | 1.15 [0.905 to 1.47]
  Toxin B IgG: Day 750: number analyzed (Participants) | 191 | 93
  Toxin B IgG: Day 750 | 2.86 [2.14 to 3.84] | 1.11 [0.840 to 1.47]
  Toxin B IgG: Day 930: number analyzed (Participants) | 108 | 66
  Toxin B IgG: Day 930 | 2.42 [1.65 to 3.55] | 1.13 [0.812 to 1.58]
  Toxin B IgG: Day 1110: number analyzed (Participants) | 59 | 36
  Toxin B IgG: Day 1110 | 3.46 [2.06 to 5.81] | 0.966 [0.592 to 1.58]

6. Secondary Outcome: Percentage of Participants With >= 2 and 4-Fold Rise in Serum Antibody Concentrations From Baseline Against Toxins A and B Measured by ELISA
Description: Percentage of Participants with >= 2 and 4-fold rise in serum antibody concentrations against toxins A and B were measured by ELISA. The 2-sided 95% Cl of the percentage was based on Exact method calculations.
Time Frame: Day 60
Population: Analysis was performed on Per Protocol Immunogenicity Analysis Set. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure and 'number analyzed' = participants with available data for each specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | C. Difficile Vaccine Group | Placebo Group
Number analyzed (Participants) | 436 | 220
percentage of participants
  Toxin A IgG: >=2: number analyzed (Participants) | 433 | 217
  Toxin A IgG: >=2 | 93.3 [90.5 to 95.5] | 0.9 [0.1 to 3.3]
  Toxin A IgG: >=4: number analyzed (Participants) | 433 | 217
  Toxin A IgG: >=4 | 88.9 [85.6 to 91.7] | 0.0 [0.0 to 1.7]
  Toxin B IgG: >=2: number analyzed (Participants) | 433 | 218
  Toxin B IgG: >=2 | 82.2 [78.3 to 85.7] | 4.6 [2.2 to 8.3]
  Toxin B IgG: >=4: number analyzed (Participants) | 433 | 218
  Toxin B IgG: >=4 | 73.2 [68.8 to 77.3] | 0.5 [0.0 to 2.5]

7. Secondary Outcome: Serum Antibody Concentrations Against Toxins A and B Measured by ELISA in Participants With CDI
Description: Serum antibody concentrations against toxins A and B were measured by ELISA and expressed as GMC. The 2-sided 95% CI GMC was based on the Student t-distribution. Symptomatic PCR-confirmed CDI cases were defined as the number of participants with combination of clinical and laboratory findings. Clinical components were: >= 3 loose stools in <= 24 hours, loose stools (defined as type 6 [fluffy pieces with ragged edges, mushy] or type 7 [watery, no solid pieces] according to the Bristol Stool Chart) lasting >= 24 hours. Laboratory findings were: stool sample positive for C. difficile Toxin B by PCR at central laboratory or diagnosis of pseudomembranous colitis visualized at colonoscopy.
Time Frame: Day 0 and Day 60
Population: Analysis was performed on participants with protocol-defined (PCR confirmed) primary CDI cases. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | C. Difficile Vaccine Group | Placebo Group
Number analyzed (Participants) | 34 | 16
EU/mL
  Toxin A IgG: Day 0: number analyzed (Participants) | 33 | 16
  Toxin A IgG: Day 0 | 1.15 [0.821 to 1.62] | 1.04 [0.661 to 1.64]
  Toxin A IgG: Day 60: number analyzed (Participants) | 30 | 16
  Toxin A IgG: Day 60 | 42.1 [18.0 to 98.3] | 1.06 [0.632 to 1.76]
  Toxin B IgG: Day 0: number analyzed (Participants) | 33 | 16
  Toxin B IgG: Day 0 | 1.41 [0.762 to 2.62] | 1.05 [0.504 to 2.20]
  Toxin B IgG: Day 60: number analyzed (Participants) | 30 | 16
  Toxin B IgG: Day 60 | 19.3 [6.65 to 56.2] | 1.13 [0.609 to 2.11]

8. Secondary Outcome: Serum Antibody Concentrations Against Toxins A and B Measured by Toxin Neutralization Assay (TNA)
Description: Serum antibody concentrations against toxins A and B were measured by TNA and expressed as geometric mean titer (GMT). The 2-sided 95% Cl of GMT was based on the Student t-distribution.
Time Frame: Day 0, Day 14, Day 30, Day 60, Day 210, Day 390, Day 570, Day 750, Day 930, and Day 1110
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titer (1/dilution)
Arm/Group | C. Difficile Vaccine Group | Placebo Group
Number analyzed (Participants) | 471 | 236
Titer (1/dilution)
  Toxin A TNA: Day 0: number analyzed (Participants) | 466 | 231
  Toxin A TNA: Day 0 | 9.86 [9.22 to 10.5] | 10.1 [9.12 to 11.2]
  Toxin A TNA: Day 14: number analyzed (Participants) | 419 | 216
  Toxin A TNA: Day 14 | 28.5 [22.7 to 35.8] | 9.86 [8.96 to 10.8]
  Toxin A TNA: Day 30: number analyzed (Participants) | 456 | 231
  Toxin A TNA: Day 30 | 50.5 [40.9 to 62.3] | 9.97 [9.09 to 10.9]
  Toxin A TNA: Day 60: number analyzed (Participants) | 416 | 212
  Toxin A TNA: Day 60 | 269 [226 to 322] | 9.82 [8.95 to 10.8]
  Toxin A TNA: Day 210: number analyzed (Participants) | 354 | 181
  Toxin A TNA: Day 210 | 269 [228 to 317] | 10.3 [9.09 to 11.7]
  Toxin A TNA: Day 390: number analyzed (Participants) | 320 | 159
  Toxin A TNA: Day 390 | 217 [183 to 259] | 10.1 [8.86 to 11.5]
  Toxin A TNA: Day 570: number analyzed (Participants) | 277 | 145
  Toxin A TNA: Day 570 | 184 [153 to 223] | 9.86 [8.76 to 11.1]
  Toxin A TNA: Day 750: number analyzed (Participants) | 191 | 93
  Toxin A TNA: Day 750 | 186 [148 to 234] | 10.2 [8.66 to 12.0]
  Toxin A TNA: Day 930: number analyzed (Participants) | 108 | 66
  Toxin A TNA: Day 930 | 173 [125 to 240] | 10.7 [8.57 to 13.4]
  Toxin A TNA: Day 1110: number analyzed (Participants) | 59 | 36
  Toxin A TNA: Day 1110 | 212 [137 to 329] | 10.2 [8.03 to 12.9]
  Toxin B TNA: Day 0: number analyzed (Participants) | 466 | 230
  Toxin B TNA: Day 0 | 12.3 [11.2 to 13.6] | 13.2 [11.2 to 15.6]
  Toxin B TNA: Day 14: number analyzed (Participants) | 419 | 216
  Toxin B TNA: Day 14 | 32.7 [25.3 to 42.2] | 13.3 [11.3 to 15.7]
  Toxin B TNA: Day 30: number analyzed (Participants) | 456 | 231
  Toxin B TNA: Day 30 | 37.8 [29.3 to 48.8] | 13.4 [11.3 to 15.8]
  Toxin B TNA: Day 60: number analyzed (Participants) | 416 | 212
  Toxin B TNA: Day 60 | 43.9 [34.0 to 56.6] | 14.3 [11.9 to 17.2]
  Toxin B TNA: Day 210: number analyzed (Participants) | 354 | 181
  Toxin B TNA: Day 210 | 41.4 [32.4 to 53.1] | 13.2 [11.1 to 15.5]
  Toxin B TNA: Day 390: number analyzed (Participants) | 319 | 159
  Toxin B TNA: Day 390 | 38.4 [30.0 to 49.0] | 13.5 [11.3 to 16.1]
  Toxin B TNA: Day 570: number analyzed (Participants) | 277 | 145
  Toxin B TNA: Day 570 | 35.7 [27.7 to 46.0] | 13.7 [11.3 to 16.8]
  Toxin B TNA: Day 750: number analyzed (Participants) | 191 | 93
  Toxin B TNA: Day 750 | 34.3 [25.1 to 46.9] | 14.6 [11.2 to 18.9]
  Toxin B TNA: Day 930: number analyzed (Participants) | 108 | 66
  Toxin B TNA: Day 930 | 31.0 [21.1 to 45.6] | 17.0 [12.3 to 23.5]
  Toxin B TNA: Day 1110: number analyzed (Participants) | 59 | 36
  Toxin B TNA: Day 1110 | 46.8 [26.1 to 84.1] | 14.0 [9.05 to 21.7]

9. Secondary Outcome: Percentage of Participants With >= 2 and 4-Fold Rise in Serum Antibody Concentrations From Baseline Against Toxins A and B Measured by TNA
Description: Percentage of Participants with >= 2 and 4-fold rise in serum antibody concentrations against toxins A and B were measured by TNA. The 2-sided 95% CI of the percentage was based on Exact method calculations.
Time Frame: Day 60
Population: Analysis was performed on Per Protocol Immunogenicity Analysis Set. Here, "overall number of participants analyzed" signifies participants evaluable for this outcome measure and 'number analyzed' = participants with evaluable data for each specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | C. Difficile Vaccine Group | Placebo Group
Number analyzed (Participants) | 436 | 220
percentage of participants
  Toxin A TNA: >=2: number analyzed (Participants) | 431 | 218
  Toxin A TNA: >=2 | 85.6 [81.9 to 88.8] | 0.5 [0.0 to 2.5]
  Toxin A TNA: >=4: number analyzed (Participants) | 431 | 218
  Toxin A TNA: >=4 | 78.2 [74.0 to 82.0] | 0.5 [0.0 to 2.5]
  Toxin B TNA: >=2: number analyzed (Participants) | 431 | 217
  Toxin B TNA: >=2 | 30.9 [26.5 to 35.5] | 2.8 [1.0 to 5.9]
  Toxin B TNA: >=4: number analyzed (Participants) | 431 | 217
  Toxin B TNA: >=4 | 27.4 [23.2 to 31.8] | 1.8 [0.5 to 4.7]

10. Secondary Outcome: Serum Antibody Concentrations Against Toxins A and B Measured by TNA in Participants With CDI
Description: Serum antibody concentrations against toxins A and B were measured by TNA and were expressed as GMT. The 2-sided 95% CI GMC was based on the Student t-distribution. Symptomatic PCR confirmed CDI cases were defined as the number of participants with combination of clinical and laboratory findings. Clinical components were: >= 3 loose stools in <= 24 hours, loose stools (defined as type 6 [fluffy pieces with ragged edges, mushy] or type 7 [watery, no solid pieces] according to the Bristol Stool Chart) lasting >= 24 hours. Laboratory findings were: stool sample positive for C. difficile Toxin B by PCR at central laboratory or diagnosis of pseudomembranous colitis visualized at colonoscopy.
Time Frame: Day 0 and Day 60
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titer (1/dilution)
Arm/Group | C. Difficile Vaccine Group | Placebo Group
Number analyzed (Participants) | 34 | 16
Titer (1/dilution)
  Toxin A TNA: Day 0: number analyzed (Participants) | 33 | 16
  Toxin A TNA: Day 0 | 12.4 [8.59 to 17.9] | 12.0 [6.27 to 23.0]
  Toxin A TNA: Day 60: number analyzed (Participants) | 30 | 16
  Toxin A TNA: Day 60 | 176 [83.4 to 371] | 10.7 [5.77 to 19.7]
  Toxin B TNA: Day 0: number analyzed (Participants) | 33 | 16
  Toxin B TNA: Day 0 | 16.7 [9.46 to 29.5] | 11.1 [7.57 to 16.3]
  Toxin B TNA: Day 60: number analyzed (Participants) | 30 | 16
  Toxin B TNA: Day 60 | 53.0 [18.3 to 153] | 13.1 [8.11 to 21.0]

11. Secondary Outcome: Percentage of Participants Reporting Solicited Injection Site and Systemic Reactions
Description: Solicited injection site reactions: pain, erythema, and swelling. Pain: Grade 1: no interference with activity, Grade 2: some interference with activity, Grade 3: significant; prevents daily activity; Erythema and swelling: Grade 1: >= 25 to <=50 mm, Grade 2: >51 to <=100 mm, Grade 3: >100 mm. Solicited systemic reactions: fever, headache, malaise, myalgia, and arthralgia. Fever: Grade 1: >= 38.0°C to <=38.4°C or >= 100.4° Fahrenheit (F) to <=101.1°F, Grade 2: >=38.5°C to <= 38.9°C or >=101.2°F to <=102.0°F, Grade 3: >=39.0°C or >=102.1°F. Headache, malaise, and myalgia: Grade 1: no interference with activity, Grade 2: some interference with activity, Grade 3: significant; prevents daily activity; Arthralgia: Grade 1: free range of motion but complains of pain or discomfort, Grade 2: decreased range of motion due to pain or discomfort, Grade 3: unwilling to move due to pain.
Time Frame: Day 0 to Day 6 after any vaccination
Population: Analysis was performed on all participants who received vaccine and were evaluable for reactogenicity. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Number; unit: percentage of participants
Arm/Group | C. Difficile Vaccine Group | Placebo Group
Number analyzed (Participants) | 1227 | 608
percentage of participants
  Injection site Pain: number analyzed (Participants) | 1199 | 586
  Injection site Pain | 38.6 | 13.5
  Injection site Erythema: number analyzed (Participants) | 1196 | 587
  Injection site Erythema | 4.2 | 0.0
  Injection site Swelling: number analyzed (Participants) | 1197 | 587
  Injection site Swelling | 3.8 | 0.3
  Fever: number analyzed (Participants) | 1173 | 577
  Fever | 4.8 | 5.7
  Headache: number analyzed (Participants) | 1196 | 586
  Headache | 25.3 | 22.5
  Malaise: number analyzed (Participants) | 1196 | 586
  Malaise | 23.9 | 19.6
  Myalgia: number analyzed (Participants) | 1196 | 586
  Myalgia | 26.6 | 21.2
  Arthralgia: number analyzed (Participants) | 1196 | 586
  Arthralgia | 19.5 | 16.7

ADVERSE EVENTS:
Time Frame: Adverse events data was collected throughout the study (up to 3 years).
Description: Safety Analysis Set included all participants who received at least one study or control vaccine and were analyzed according to the vaccine received. Solicited reaction(SR) was an adverse event (AE) that was prelisted (i.e.,solicited) in the electronic case report form (eCRF) and considered to be related to vaccination. An unsolicited AE was an observed AE that did not fulfill the conditions prelisted (i.e.,solicited) in the eCRF in terms of symptom and/or onset post-vaccination.
Arm/Group | C. Difficile Vaccine Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 255/6113 | 127/3057
Serious Adverse Events (participants affected / at risk) | 1662/6113 | 851/3057
Other Adverse Events (participants affected / at risk) | 1347/6113 | 401/3057
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | C. Difficile Vaccine Group (N=6113) | Placebo Group (N=3057)
Anaemia (Blood and lymphatic system disorders) | 19 (20) | 11 (13)
Antiphospholipid Syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Haemolytic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 2 (2) | 5 (5)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Microcytic Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Nephrogenic Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Normochromic Normocytic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute Coronary Syndrome (Cardiac disorders) | 13 (15) | 2 (2)
Acute Myocardial Infarction (Cardiac disorders) | 56 (59) | 22 (24)
Angina Pectoris (Cardiac disorders) | 19 (20) | 10 (10)
Angina Unstable (Cardiac disorders) | 27 (32) | 9 (15)
Aortic Valve Incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Aortic Valve Stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 9 (9) | 2 (2)
Arrhythmia Supraventricular (Cardiac disorders) | 2 (2) | 0 (0)
Arteriosclerosis Coronary Artery (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 42 (53) | 14 (15)
Atrial Flutter (Cardiac disorders) | 3 (3) | 2 (2)
Atrial Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Atrial Thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular Block (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular Block Complete (Cardiac disorders) | 0 (0) | 2 (2)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 5 (6) | 5 (5)
Bundle Branch Block Left (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 10 (11) | 8 (8)
Cardiac Disorder (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac Failure (Cardiac disorders) | 34 (40) | 16 (36)
Cardiac Failure Acute (Cardiac disorders) | 16 (22) | 6 (7)
Cardiac Failure Chronic (Cardiac disorders) | 3 (5) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 69 (102) | 29 (37)
Cardiac Tamponade (Cardiac disorders) | 6 (6) | 2 (2)
Cardiac Valve Disease (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-Respiratory Arrest (Cardiac disorders) | 10 (11) | 3 (3)
Cardiogenic Shock (Cardiac disorders) | 8 (9) | 5 (5)
Cardiomyopathy (Cardiac disorders) | 5 (6) | 1 (1)
Cardiopulmonary Failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiorenal Syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Cor Pulmonale (Cardiac disorders) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 22 (23) | 7 (7)
Coronary Artery Occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Coronary Artery Stenosis (Cardiac disorders) | 7 (8) | 2 (2)
Coronary Artery Thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Heart Valve Incompetence (Cardiac disorders) | 1 (1) | 1 (1)
Hypertensive Heart Disease (Cardiac disorders) | 1 (1) | 0 (0)
Intracardiac Thrombus (Cardiac disorders) | 1 (1) | 2 (2)
Ischaemic Cardiomyopathy (Cardiac disorders) | 1 (1) | 2 (2)
Left Ventricular Failure (Cardiac disorders) | 1 (1) | 0 (0)
Mitral Valve Incompetence (Cardiac disorders) | 3 (3) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 27 (27) | 16 (16)
Myocardial Ischaemia (Cardiac disorders) | 8 (8) | 3 (3)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 5 (5) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 2 (2)
Prinzmetal Angina (Cardiac disorders) | 1 (1) | 0 (0)
Pulseless Electrical Activity (Cardiac disorders) | 0 (0) | 1 (1)
Reperfusion Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Right Ventricular Failure (Cardiac disorders) | 1 (1) | 0 (0)
Sick Sinus Syndrome (Cardiac disorders) | 2 (2) | 3 (3)
Sinoatrial Block (Cardiac disorders) | 1 (1) | 0 (0)
Sinus Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Stress Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Tricuspid Valve Incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Ventricle Rupture (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Fibrillation (Cardiac disorders) | 3 (3) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 5 (5) | 4 (4)
Anophthalmos (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Cardiac Septal Defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Ectopic Ureter (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Deafness Neurosensory (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Meniere's Disease (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Sudden Hearing Loss (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Vertigo Positional (Ear and labyrinth disorders) | 4 (4) | 0 (0)
Adrenal Insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hyperparathyroidism Primary (Endocrine disorders) | 1 (1) | 0 (0)
Thyroid Mass (Endocrine disorders) | 2 (2) | 1 (1)
Amaurosis (Eye disorders) | 1 (1) | 1 (1)
Amaurosis Fugax (Eye disorders) | 2 (2) | 0 (0)
Aphakia (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 2 (2) | 2 (3)
Conjunctivochalasis (Eye disorders) | 1 (1) | 0 (0)
Eyelid Ptosis (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Phacolytic Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Pterygium (Eye disorders) | 1 (1) | 0 (0)
Retinal Detachment (Eye disorders) | 0 (0) | 1 (1)
Retinal Vein Occlusion (Eye disorders) | 1 (1) | 0 (0)
Vitreous Haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Abdominal Adhesions (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal Hernia (Gastrointestinal disorders) | 3 (3) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 14 (14) | 11 (15)
Abdominal Pain Lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal Wall Haematoma (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anal Fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal Fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Change Of Bowel Habit (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 5 (5) | 0 (0)
Colitis Ischaemic (Gastrointestinal disorders) | 1 (1) | 2 (2)
Colitis Microscopic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic Pseudo-Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic Stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 9 (9) | 2 (2)
Crohn's Disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dental Pulp Disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diabetic Gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diaphragmatic Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 2 (2)
Diverticular Perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 4 (5) | 1 (1)
Duodenal Ulcer (Gastrointestinal disorders) | 2 (2) | 1 (1)
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterovesical Fistula (Gastrointestinal disorders) | 1 (2) | 1 (1)
Erosive Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Erosive Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food Poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric Disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric Haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastric Ulcer (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric Ulcer Perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 8 (8) | 4 (5)
Gastritis Erosive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis Haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroduodenal Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Amyloidosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 13 (13) | 6 (6)
Gastrointestinal Hypomotility (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hernial Eventration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus Hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ileal Stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 6 (6) | 2 (2)
Ileus Paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired Gastric Emptying (Gastrointestinal disorders) | 1 (5) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 4 (4) | 3 (3)
Inguinal Hernia, Obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 6 (7) | 1 (1)
Intestinal Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-Abdominal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large Intestine Polyp (Gastrointestinal disorders) | 5 (5) | 0 (0)
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 4 (4) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 2 (2)
Mesenteric Artery Thrombosis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Mesenteric Vein Thrombosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Oesophageal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal Stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal Varices Haemorrhage (Gastrointestinal disorders) | 2 (3) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral Disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic Pseudocyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 6 (7) | 3 (3)
Pancreatitis Acute (Gastrointestinal disorders) | 4 (5) | 6 (6)
Pancreatitis Chronic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis Relapsing (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic Ulcer (Gastrointestinal disorders) | 1 (1) | 2 (2)
Periodontal Disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritoneal Adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritoneal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal Haemorrhage (Gastrointestinal disorders) | 4 (4) | 2 (2)
Rectal Prolapse (Gastrointestinal disorders) | 2 (2) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 5 (5) | 2 (2)
Spigelian Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Thrombosis Mesenteric Vessel (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical Hernia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Umbilical Hernia, Obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 5 (5) | 2 (2)
Varices Oesophageal (Gastrointestinal disorders) | 2 (2) | 0 (0)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 2 (2)
Asthenia (General disorders) | 4 (4) | 2 (2)
Catheter Site Haemorrhage (General disorders) | 2 (2) | 0 (0)
Chest Discomfort (General disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 50 (56) | 19 (27)
Death (General disorders) | 8 (8) | 6 (6)
Device Dislocation (General disorders) | 9 (9) | 1 (1)
Device Failure (General disorders) | 3 (3) | 2 (2)
Device Issue (General disorders) | 1 (1) | 0 (0)
Device Leakage (General disorders) | 1 (1) | 0 (0)
Device Malfunction (General disorders) | 1 (1) | 1 (1)
Device Occlusion (General disorders) | 2 (2) | 1 (1)
Drug Interaction (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
General Physical Health Deterioration (General disorders) | 1 (1) | 1 (1)
General Symptom (General disorders) | 1 (1) | 0 (0)
Generalised Oedema (General disorders) | 0 (0) | 1 (1)
Hernia Obstructive (General disorders) | 0 (0) | 1 (1)
Hyperthermia (General disorders) | 1 (1) | 0 (0)
Impaired Healing (General disorders) | 1 (1) | 0 (0)
Implant Site Haematoma (General disorders) | 1 (1) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 1 (1)
Medical Device Complication (General disorders) | 7 (8) | 4 (4)
Multi-Organ Failure (General disorders) | 4 (4) | 3 (3)
Non-Cardiac Chest Pain (General disorders) | 2 (2) | 2 (2)
Oedema (General disorders) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 3 (3) | 1 (1)
Pain (General disorders) | 2 (2) | 3 (3)
Patient-Device Incompatibility (General disorders) | 0 (0) | 1 (1)
Perforated Ulcer (General disorders) | 1 (1) | 0 (0)
Polyp (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 5 (5) | 3 (3)
Spinal Pain (General disorders) | 1 (1) | 0 (0)
Stent-Graft Endoleak (General disorders) | 1 (1) | 1 (1)
Sudden Cardiac Death (General disorders) | 2 (2) | 1 (1)
Sudden Death (General disorders) | 2 (2) | 1 (1)
Surgical Failure (General disorders) | 0 (0) | 1 (1)
Systemic Inflammatory Response Syndrome (General disorders) | 1 (1) | 2 (2)
Bile Duct Obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile Duct Stenosis (Hepatobiliary disorders) | 1 (2) | 0 (0)
Bile Duct Stone (Hepatobiliary disorders) | 3 (3) | 3 (3)
Cholangitis (Hepatobiliary disorders) | 2 (2) | 3 (3)
Cholangitis Acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 7 (7) | 1 (1)
Cholecystitis Acute (Hepatobiliary disorders) | 2 (2) | 7 (7)
Cholecystitis Chronic (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 7 (7) | 6 (6)
Cirrhosis Alcoholic (Hepatobiliary disorders) | 2 (2) | 1 (2)
Gallbladder Polyp (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic Cirrhosis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Hepatic Cyst (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic Failure (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis Acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatorenal Syndrome (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hydrocholecystis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic Reaction (Immune system disorders) | 2 (2) | 0 (0)
Anaphylactic Shock (Immune system disorders) | 1 (1) | 0 (0)
Device Allergy (Immune system disorders) | 1 (1) | 0 (0)
Food Allergy (Immune system disorders) | 1 (1) | 0 (0)
Secondary Immunodeficiency (Immune system disorders) | 0 (0) | 1 (1)
Abdominal Hernia Gangrenous (Infections and infestations) | 1 (1) | 0 (0)
Abdominal Infection (Infections and infestations) | 1 (1) | 0 (0)
Abdominal Sepsis (Infections and infestations) | 2 (2) | 3 (3)
Abdominal Wall Abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 4 (5) | 0 (0)
Abscess Limb (Infections and infestations) | 4 (4) | 2 (2)
Anal Abscess (Infections and infestations) | 2 (2) | 1 (1)
Appendicitis (Infections and infestations) | 5 (5) | 2 (2)
Appendicitis Perforated (Infections and infestations) | 1 (1) | 0 (0)
Arteriovenous Graft Site Abscess (Infections and infestations) | 1 (1) | 0 (0)
Arthritis Bacterial (Infections and infestations) | 11 (11) | 3 (3)
Arthritis Infective (Infections and infestations) | 8 (9) | 3 (4)
Asymptomatic Bacteriuria (Infections and infestations) | 1 (1) | 0 (0)
Atypical Mycobacterial Infection (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 8 (9) | 2 (2)
Bacterial Infection (Infections and infestations) | 1 (1) | 1 (1)
Bacterial Sepsis (Infections and infestations) | 4 (4) | 0 (0)
Bacterial Tracheitis (Infections and infestations) | 0 (0) | 1 (1)
Beta Haemolytic Streptococcal Infection (Infections and infestations) | 1 (1) | 1 (1)
Biliary Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Breast Abscess (Infections and infestations) | 1 (1) | 0 (0)
Breast Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 11 (11) | 3 (3)
Bronchopneumonia (Infections and infestations) | 3 (3) | 0 (0)
Bursitis Infective (Infections and infestations) | 1 (1) | 0 (0)
Candida Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 63 (78) | 36 (41)
Chronic Hepatitis C (Infections and infestations) | 0 (0) | 1 (1)
Clostridium Difficile Colitis (Infections and infestations) | 3 (3) | 0 (0)
Clostridium Difficile Infection (Infections and infestations) | 3 (3) | 1 (1)
Dengue Fever (Infections and infestations) | 2 (2) | 2 (2)
Dermo-Hypodermitis (Infections and infestations) | 1 (1) | 0 (0)
Device Related Infection (Infections and infestations) | 18 (22) | 12 (14)
Diabetic Foot Infection (Infections and infestations) | 26 (30) | 9 (9)
Diabetic Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea Infectious (Infections and infestations) | 1 (1) | 0 (0)
Disseminated Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 4 (4) | 2 (2)
Empyema (Infections and infestations) | 0 (0) | 2 (2)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis Infectious (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 3 (3) | 1 (1)
Escherichia Bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
Escherichia Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia Urinary Tract Infection (Infections and infestations) | 2 (2) | 0 (0)
Gangrene (Infections and infestations) | 2 (2) | 1 (3)
Gastric Infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 10 (10) | 6 (6)
Gastroenteritis Viral (Infections and infestations) | 3 (3) | 0 (0)
Genital Herpes (Infections and infestations) | 1 (1) | 0 (0)
Graft Infection (Infections and infestations) | 2 (2) | 0 (0)
Groin Abscess (Infections and infestations) | 3 (3) | 0 (0)
Haematoma Infection (Infections and infestations) | 1 (1) | 0 (0)
Hepatic Cyst Infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes Virus Infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes Zoster (Infections and infestations) | 3 (3) | 1 (1)
Implant Site Infection (Infections and infestations) | 2 (2) | 0 (0)
Incision Site Infection (Infections and infestations) | 0 (0) | 1 (1)
Infected Skin Ulcer (Infections and infestations) | 2 (3) | 2 (2)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Infection In An Immunocompromised Host (Infections and infestations) | 1 (1) | 0 (0)
Infective Exacerbation Of Bronchiectasis (Infections and infestations) | 2 (6) | 0 (0)
Infective Exacerbation Of Chronic Obstructive Airways Disease (Infections and infestations) | 2 (2) | 1 (1)
Infective Spondylitis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 5 (5) | 2 (2)
Intervertebral Discitis (Infections and infestations) | 3 (3) | 0 (0)
Joint Abscess (Infections and infestations) | 1 (1) | 0 (0)
Kidney Infection (Infections and infestations) | 1 (1) | 0 (0)
Liver Abscess (Infections and infestations) | 1 (1) | 1 (1)
Lobar Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Localised Infection (Infections and infestations) | 4 (4) | 4 (5)
Lower Respiratory Tract Infection (Infections and infestations) | 7 (7) | 2 (2)
Lower Respiratory Tract Infection Viral (Infections and infestations) | 1 (1) | 0 (0)
Lung Infection (Infections and infestations) | 1 (1) | 1 (1)
Mediastinitis (Infections and infestations) | 4 (4) | 2 (2)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Mumps (Infections and infestations) | 1 (1) | 0 (0)
Mycobacterium Avium Complex Infection (Infections and infestations) | 0 (0) | 1 (1)
Nail Infection (Infections and infestations) | 1 (1) | 0 (0)
Neurological Infection (Infections and infestations) | 0 (0) | 1 (1)
Neurosyphilis (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 6 (6) | 1 (2)
Osteomyelitis (Infections and infestations) | 27 (29) | 11 (16)
Osteomyelitis Acute (Infections and infestations) | 2 (2) | 0 (0)
Osteomyelitis Chronic (Infections and infestations) | 2 (2) | 2 (2)
Otitis Externa (Infections and infestations) | 1 (1) | 0 (0)
Paraspinal Abscess (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Perihepatic Abscess (Infections and infestations) | 1 (1) | 0 (0)
Perineal Abscess (Infections and infestations) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 2 (2) | 0 (0)
Peritonitis (Infections and infestations) | 2 (2) | 0 (0)
Peritonsillar Abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 107 (122) | 67 (84)
Pneumonia Bacterial (Infections and infestations) | 5 (9) | 2 (2)
Pneumonia Necrotising (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia Pneumococcal (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia Staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Poliomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Post Procedural Cellulitis (Infections and infestations) | 1 (1) | 1 (2)
Post Procedural Infection (Infections and infestations) | 7 (7) | 1 (1)
Post Procedural Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Post Procedural Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Postoperative Wound Infection (Infections and infestations) | 28 (30) | 15 (15)
Prostatic Abscess (Infections and infestations) | 1 (1) | 0 (0)
Psoas Abscess (Infections and infestations) | 0 (0) | 2 (2)
Pulmonary Sepsis (Infections and infestations) | 1 (2) | 2 (2)
Pulmonary Tuberculosis (Infections and infestations) | 2 (2) | 0 (0)
Pyelonephritis (Infections and infestations) | 5 (5) | 2 (2)
Pyelonephritis Acute (Infections and infestations) | 7 (8) | 1 (1)
Renal Abscess (Infections and infestations) | 1 (1) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 7 (8) | 4 (6)
Scrotal Abscess (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 34 (38) | 18 (18)
Septic Arthritis Staphylococcal (Infections and infestations) | 2 (2) | 0 (0)
Septic Shock (Infections and infestations) | 26 (27) | 13 (13)
Sinusitis Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Skin Bacterial Infection (Infections and infestations) | 3 (4) | 0 (0)
Skin Infection (Infections and infestations) | 2 (2) | 2 (2)
Soft Tissue Infection (Infections and infestations) | 3 (3) | 4 (4)
Staphylococcal Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal Infection (Infections and infestations) | 4 (4) | 3 (3)
Staphylococcal Osteomyelitis (Infections and infestations) | 1 (1) | 2 (2)
Staphylococcal Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Subcutaneous Abscess (Infections and infestations) | 0 (0) | 2 (2)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 2 (2) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary Bladder Abscess (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 91 (116) | 38 (47)
Urinary Tract Infection Bacterial (Infections and infestations) | 3 (3) | 1 (1)
Urinary Tract Infection Pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 11 (12) | 6 (6)
Viral Infection (Infections and infestations) | 0 (0) | 1 (1)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Wound Infection (Infections and infestations) | 5 (5) | 1 (1)
Wound Infection Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Abdominal Wound Dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Accidental Overdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Alcohol Poisoning (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Anaemia Postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Animal Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle Fracture (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Arterial Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bladder Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bone Fissure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac Procedure Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chemical Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Coronary Artery Restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Dislocation Of Vertebra (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dural Tear (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Exposure To Toxic Agent (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Extradural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 17 (18) | 7 (7)
Fat Embolism (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Femur Fracture (Injury, poisoning and procedural complications) | 11 (12) | 4 (4)
Foot Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Forearm Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Heat Exhaustion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Heat Stroke (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 8 (8) | 6 (7)
Humerus Fracture (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Incisional Hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint Dislocation (Injury, poisoning and procedural complications) | 12 (16) | 0 (0)
Joint Dislocation Postoperative (Injury, poisoning and procedural complications) | 4 (5) | 0 (0)
Joint Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament Injury (Injury, poisoning and procedural complications) | 2 (3) | 1 (1)
Ligament Rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament Sprain (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Mechanical Ventilation Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus Injury (Injury, poisoning and procedural complications) | 0 (0) | 5 (6)
Multiple Fractures (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Multiple Injuries (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Muscle Rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle Strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Patella Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Pelvic Fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Periprosthetic Fracture (Injury, poisoning and procedural complications) | 6 (7) | 5 (6)
Pneumothorax Traumatic (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post Concussion Syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post Procedural Complication (Injury, poisoning and procedural complications) | 18 (18) | 11 (13)
Post Procedural Discharge (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post Procedural Haematuria (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Post Procedural Swelling (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative Fever (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Postoperative Ileus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative Respiratory Failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative Thoracic Procedure Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative Wound Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural Haemorrhage (Injury, poisoning and procedural complications) | 4 (5) | 0 (0)
Procedural Hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural Nausea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Pubis Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rectal Laceration Postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Renal Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Road Traffic Accident (Injury, poisoning and procedural complications) | 2 (2) | 5 (5)
Scrotal Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Spinal Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Stab Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stress Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural Haematoma (Injury, poisoning and procedural complications) | 6 (6) | 3 (3)
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon Rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal Burn (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Tibia Fracture (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Tracheostomy Malfunction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Traumatic Arthritis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic Intracranial Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urethral Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urethral Stricture Postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular Bypass Dysfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular Graft Occlusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Vascular Graft Thrombosis (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound Dehiscence (Injury, poisoning and procedural complications) | 3 (5) | 2 (2)
Wrist Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anticoagulation Drug Level Above Therapeutic (Investigations) | 0 (0) | 1 (1)
Aspiration Bronchial (Investigations) | 1 (1) | 0 (0)
Blood Creatinine Increased (Investigations) | 1 (1) | 0 (0)
Blood Potassium Decreased (Investigations) | 0 (0) | 1 (1)
Carbon Dioxide Abnormal (Investigations) | 1 (1) | 0 (0)
Cardiac Pacemaker Evaluation (Investigations) | 1 (1) | 0 (0)
Coagulation Time Prolonged (Investigations) | 0 (0) | 1 (1)
Electrocardiogram St Segment Elevation (Investigations) | 1 (1) | 0 (0)
Influenza A Virus Test Positive (Investigations) | 1 (1) | 0 (0)
International Normalised Ratio Increased (Investigations) | 1 (1) | 0 (0)
Oxygen Saturation Decreased (Investigations) | 0 (0) | 1 (1)
Prothrombin Time Abnormal (Investigations) | 1 (1) | 0 (0)
Transaminases Increased (Investigations) | 0 (0) | 1 (1)
Urine Output Decreased (Investigations) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Central Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
Diabetes Mellitus (Metabolism and nutrition disorders) | 12 (15) | 2 (2)
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 8 (11) | 2 (2)
Diabetic Complication (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 3 (4) | 2 (2)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Fluid Overload (Metabolism and nutrition disorders) | 4 (6) | 5 (13)
Gout (Metabolism and nutrition disorders) | 5 (6) | 0 (0)
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 10 (12) | 6 (6)
Hyperglycaemic Hyperosmolar Nonketotic Syndrome (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (6) | 4 (4)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 11 (11) | 6 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (6) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Obesity (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Type 1 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Ankylosing Spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (10) | 4 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 8 (10)
Bursitis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chronic Recurrent Multifocal Osteomyelitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Collagen Disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Foot Deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fracture Nonunion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Gouty Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Joint Instability (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle Necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 47 (51) | 19 (19)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (3)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Abdominal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Adenocarcinoma Gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Adenocarcinoma Of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adrenal Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Benign Bone Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Bladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Bladder Transitional Cell Carcinoma Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder Transitional Cell Carcinoma Stage Ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bone Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Brain Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Breast Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Breast Cancer Stage Ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Burkitt's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoid Tumour Of The Duodenum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervix Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cervix Carcinoma Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0)
Cervix Carcinoma Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Clear Cell Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 1 (1)
Colon Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Diffuse Large B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Endometrial Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Eyelid Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gallbladder Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Gastric Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal Stromal Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Glioblastoma Multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Intraductal Papillary Mucinous Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Kaposi's Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung Carcinoma Cell Type Unspecified Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung Carcinoma Cell Type Unspecified Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant Neoplasm Of Eye (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant Neoplasm Of Renal Pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant Pleural Effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant Respiratory Tract Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mantle Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mediastinum Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases To Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic Carcinoma Of The Bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 0 (0)
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Neoplasm Of Thymus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm Prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroendocrine Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Nodal Marginal Zone B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Non-Small Cell Lung Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (4) | 0 (0)
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Ovarian Epithelial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Pancreatic Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic Neuroendocrine Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Parathyroid Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Plasma Cell Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 17 (17) | 3 (3)
Prostate Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Renal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Retroperitoneal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Salivary Gland Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Salivary Gland Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small Intestine Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Superficial Spreading Melanoma Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Testicular Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Altered State Of Consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Apallic Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Arachnoid Cyst (Nervous system disorders) | 1 (1) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Brain Stem Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Carotid Arteriosclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Carotid Artery Stenosis (Nervous system disorders) | 2 (2) | 1 (1)
Carpal Tunnel Syndrome (Nervous system disorders) | 0 (0) | 2 (2)
Cerebral Artery Stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral Haemorrhage (Nervous system disorders) | 4 (4) | 2 (2)
Cerebral Infarction (Nervous system disorders) | 5 (5) | 7 (7)
Cerebral Ischaemia (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral Thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 19 (20) | 8 (8)
Cerebrovascular Disorder (Nervous system disorders) | 3 (3) | 3 (3)
Cervical Myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Cervicobrachial Syndrome (Nervous system disorders) | 0 (0) | 2 (2)
Chronic Inflammatory Demyelinating Polyradiculoneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 11 (15) | 9 (22)
Critical Illness Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Dementia Alzheimer's Type (Nervous system disorders) | 0 (0) | 1 (1)
Dementia With Lewy Bodies (Nervous system disorders) | 1 (1) | 1 (1)
Diabetic Neuropathy (Nervous system disorders) | 0 (0) | 2 (3)
Dizziness (Nervous system disorders) | 4 (4) | 4 (4)
Dizziness Postural (Nervous system disorders) | 1 (1) | 0 (0)
Embolic Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 5 (5) | 4 (4)
Epilepsy (Nervous system disorders) | 2 (3) | 1 (3)
Facial Paresis (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage Intracranial (Nervous system disorders) | 1 (1) | 1 (1)
Haemorrhagic Stroke (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 2 (2)
Hemiplegic Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Hepatic Encephalopathy (Nervous system disorders) | 2 (6) | 4 (7)
Hydrocephalus (Nervous system disorders) | 1 (1) | 1 (2)
Hypertensive Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycaemic Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hypoxic-Ischaemic Encephalopathy (Nervous system disorders) | 3 (3) | 1 (1)
Intercostal Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial Aneurysm (Nervous system disorders) | 1 (1) | 2 (2)
Intracranial Pressure Increased (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic Cerebral Infarction (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic Stroke (Nervous system disorders) | 11 (13) | 5 (5)
Lacunar Infarction (Nervous system disorders) | 1 (1) | 0 (0)
Lumbar Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 3 (3) | 1 (1)
Neuropathy Peripheral (Nervous system disorders) | 0 (0) | 2 (2)
Normal Pressure Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Partial Seizures (Nervous system disorders) | 1 (2) | 0 (0)
Pneumocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Post-Traumatic Headache (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 3 (3) | 1 (1)
Radicular Pain (Nervous system disorders) | 1 (1) | 0 (0)
Radicular Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Spinal Cord Compression (Nervous system disorders) | 0 (0) | 1 (1)
Status Epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid Haemorrhage (Nervous system disorders) | 3 (3) | 0 (0)
Syncope (Nervous system disorders) | 14 (15) | 9 (9)
Tension Headache (Nervous system disorders) | 0 (0) | 1 (1)
Thalamus Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Toxic Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Transient Global Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 21 (21) | 8 (8)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Trigeminal Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Vertebrobasilar Insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Vertigo Cns Origin (Nervous system disorders) | 0 (0) | 1 (1)
Vocal Cord Paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Alcohol Abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 2 (3) | 0 (0)
Completed Suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Conversion Disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Delirium (Psychiatric disorders) | 2 (2) | 4 (4)
Depression (Psychiatric disorders) | 4 (5) | 1 (1)
Drug Dependence (Psychiatric disorders) | 1 (1) | 0 (0)
Impaired Self-Care (Psychiatric disorders) | 1 (1) | 0 (0)
Major Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Mental Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 4 (4) | 5 (5)
Panic Attack (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Schizoaffective Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Schizophrenia (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 3 (3)
Suicide Attempt (Psychiatric disorders) | 1 (1) | 1 (1)
Azotaemia (Renal and urinary disorders) | 2 (2) | 0 (0)
Bladder Mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder Neck Obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder Outlet Obstruction (Renal and urinary disorders) | 2 (2) | 0 (0)
Calculus Ureteric (Renal and urinary disorders) | 2 (2) | 2 (3)
Calculus Urinary (Renal and urinary disorders) | 2 (2) | 0 (0)
Cystitis Interstitial (Renal and urinary disorders) | 0 (0) | 1 (1)
Diabetic Nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 8 (8) | 6 (7)
Hydronephrosis (Renal and urinary disorders) | 4 (4) | 0 (0)
Lupus Nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Micturition Disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 9 (10) | 1 (2)
Nephrotic Syndrome (Renal and urinary disorders) | 0 (0) | 1 (1)
Obstructive Uropathy (Renal and urinary disorders) | 2 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 7 (8) | 3 (3)
Renal Failure Acute (Renal and urinary disorders) | 31 (35) | 8 (9)
Renal Failure Chronic (Renal and urinary disorders) | 17 (19) | 3 (3)
Renal Haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Impairment (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Tubular Necrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Strangury (Renal and urinary disorders) | 1 (1) | 0 (0)
Stress Urinary Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Tubulointerstitial Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureteric Stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral Stenosis (Renal and urinary disorders) | 7 (8) | 6 (9)
Urinary Incontinence (Renal and urinary disorders) | 3 (5) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 5 (8) | 2 (2)
Urinoma (Renal and urinary disorders) | 0 (0) | 1 (1)
Vesicocutaneous Fistula (Renal and urinary disorders) | 0 (0) | 1 (2)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 8 (8) | 5 (5)
Breast Enlargement (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Epididymitis (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Female Genital Tract Fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Genital Prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian Cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Postmenopausal Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine Haemorrhage (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal Prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 23 (29) | 10 (12)
Alveolitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 18 (23) | 3 (4)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 84 (121) | 51 (71)
Chronic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 (15) | 15 (15)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (5)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Idiopathic Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 1 (1)
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung Hernia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Mediastinal Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Mediastinal Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Obstructive Airways Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 21 (22) | 10 (11)
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 1 (1)
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 23 (23) | 17 (17)
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary Microemboli (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 16 (18) | 12 (15)
Sinus Polyp (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3)
Status Asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tracheal Stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetic Foot (Skin and subcutaneous tissue disorders) | 24 (25) | 13 (14)
Diabetic Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 11 (12) | 7 (9)
Stevens-Johnson Syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Artificial Urinary Sphincter Implant (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac Pacemaker Battery Replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardioversion (Surgical and medical procedures) | 0 (0) | 1 (1)
Cerebrospinal Fluid Drainage (Surgical and medical procedures) | 0 (0) | 1 (1)
Hip Arthroplasty (Surgical and medical procedures) | 1 (1) | 1 (1)
Incisional Drainage (Surgical and medical procedures) | 0 (0) | 1 (1)
Knee Arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee Operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Leg Amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Metatarsal Excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Parathyroidectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Rehabilitation Therapy (Surgical and medical procedures) | 2 (2) | 0 (0)
Tooth Extraction (Surgical and medical procedures) | 1 (1) | 0 (0)
Aneurysm (Vascular disorders) | 0 (0) | 1 (2)
Aneurysm Ruptured (Vascular disorders) | 1 (1) | 0 (0)
Aortic Aneurysm (Vascular disorders) | 1 (1) | 3 (3)
Aortic Aneurysm Rupture (Vascular disorders) | 0 (0) | 1 (1)
Aortic Stenosis (Vascular disorders) | 2 (2) | 2 (2)
Aortic Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Arterial Occlusive Disease (Vascular disorders) | 2 (2) | 1 (1)
Arterial Stenosis (Vascular disorders) | 2 (2) | 0 (0)
Arteriosclerosis (Vascular disorders) | 4 (4) | 0 (0)
Circulatory Collapse (Vascular disorders) | 1 (2) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 12 (12) | 5 (5)
Essential Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Extremity Necrosis (Vascular disorders) | 2 (2) | 0 (0)
Femoral Artery Occlusion (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 4 (4) | 2 (2)
Hypertension (Vascular disorders) | 7 (7) | 2 (2)
Hypertensive Crisis (Vascular disorders) | 9 (9) | 1 (1)
Hypertensive Emergency (Vascular disorders) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 5 (5)
Hypovolaemic Shock (Vascular disorders) | 4 (4) | 4 (4)
Infarction (Vascular disorders) | 0 (0) | 1 (1)
Intra-Abdominal Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1) | 1 (1)
Orthostatic Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 7 (8) | 4 (4)
Peripheral Artery Aneurysm (Vascular disorders) | 0 (0) | 1 (2)
Peripheral Artery Stenosis (Vascular disorders) | 4 (5) | 0 (0)
Peripheral Artery Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Embolism (Vascular disorders) | 0 (0) | 1 (1)
Peripheral Ischaemia (Vascular disorders) | 11 (15) | 1 (1)
Peripheral Vascular Disorder (Vascular disorders) | 12 (13) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 1 (1)
Phlebitis Deep (Vascular disorders) | 0 (0) | 1 (1)
Post Thrombotic Syndrome (Vascular disorders) | 1 (2) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 1 (1)
Shock Haemorrhagic (Vascular disorders) | 5 (5) | 1 (1)
Subclavian Artery Stenosis (Vascular disorders) | 0 (0) | 1 (1)
Temporal Arteritis (Vascular disorders) | 1 (1) | 0 (0)
Thromboangiitis Obliterans (Vascular disorders) | 1 (2) | 0 (0)
Thrombophlebitis Superficial (Vascular disorders) | 1 (2) | 0 (0)
Varicophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Varicose Ulceration (Vascular disorders) | 1 (1) | 2 (2)
Vascular Insufficiency (Vascular disorders) | 1 (1) | 0 (0)
Venous Thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Venous Thrombosis Limb (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | C. Difficile Vaccine Group (N=6113) | Placebo Group (N=3057)
Injection Site Pain (General disorders) | 855 (1252) | 127 (157)
Malaise (General disorders) | 325 (456) | 135 (195)
Arthralgia (Musculoskeletal and connective tissue disorders) | 345 (481) | 146 (205)
Myalgia (Musculoskeletal and connective tissue disorders) | 368 (556) | 132 (201)
Headache (Nervous system disorders) | 531 (758) | 229 (327)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2017-02-14): https://cdn.clinicaltrials.gov/large-docs/12/NCT01887912/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-05): https://cdn.clinicaltrials.gov/large-docs/12/NCT01887912/SAP_001.pdf